CLINICAL TRIAL: NCT04685876
Title: Comparison of Liposomal Bupivacaine, Plain Bupivacaine, and Placebo for Transversus Abdominis Plane Blocks: A Randomized, Blinded Trial
Brief Title: Comparing TAP Blocks Bupivacaine, and Placebo for Plane
Acronym: CLEVELAND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Edward Mascha (Other)
Responsible Party: Sponsor-Investigator, Edward Mascha, PhD, Staff, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20-790
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Abdominal Surgery
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- liposomal bupivacaine (Active Comparator): 40 ml of plain bupivacaine 0.25% will be mixed with 20 ml liposomal bupivacaine and 20 ml of saline. 20 ml of the mix will be injected at each location of the 4-quadrant TAP block.
  Interventions: Drug: Liposomal bupivacaine
- plain bupivacaine (Active Comparator): 50 ml of plain bupivacaine 0.5% will be combined with 30 ml of normal saline making a total of 80 ml. 20 ml will be injected at each location of the 4-quadrant TAP block.
  Interventions: Drug: Plain bupivacaine
- Normal Saline (Placebo Comparator): patients will receive total of 80 ml of normal saline, injected 20 ml in each of the four-quadrant sites.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Liposomal bupivacaine — 4-quadrant TAP block with liposomal bupivacaine
  Arms: liposomal bupivacaine
Drug: Plain bupivacaine — 4-quadrant TAP block with plain bupivacaine
  Arms: plain bupivacaine
Drug: Normal saline — placebo (normal saline).
  Arms: Normal Saline

SUMMARY:
The study will prospectively compare the analgesic efficacy of TAP blocks with liposomal bupivacaine, plain bupivacaine, and placebo in patients who are scheduled for major abdominal surgery. The primary aim is to assess the duration of the local analgesia (determined by pinprick and cold) in all four quadrants. Comparing opioid consumption and pain scores is a secondary aim. All aims will be assessed over 72 hours or the duration of hospitalization if shorter.

DETAILED DESCRIPTION:
The investigators propose a randomized double-blind trial comparing TAP blocks with liposomal bupivacaine, plain bupivacaine, and placebo in patients having elective abdominal surgery.

After eligibility is confirmed, patients will receive complete information about the study both verbally and in writing. Informed consent will be obtained from the patients prior to randomization and study-specific procedures.

Randomization will be based on computer-generated codes and use random-sized blocks. Allocations will be concealed until the morning of surgery where they will be provided by a web-based system. Randomization will be stratified by study site and chronic opioid use, defined by opioid use for more than 30 consecutive days within three preoperative months, at a daily dose of 15 mg or more of morphine or equivalent. Randomization will also be stratified according to anticipated type of surgery (open vs. laparoscopic-assisted). Clinicians doing the blocks will not be involved in data collection and all the evaluators will be blinded to group allocations.

All blocks will be performed preoperatively or after induction of anesthesia by attending anesthesiologists or regional anesthesia fellows who are experienced in TAP blocks. Premedication will be administered at the discretion of the attending anesthesiologist and standard monitors will be used. Patients will be given 1 g oral acetaminophen an hour before surgery, and an additional 500 mg every 6 hours for 72 hours after surgery starting with oral intake.

Patients will be randomly assigned to: 1) 4-quadrant TAP block with liposomal bupivacaine; 2) 4-quadrant TAP block with plain bupivacaine; or, 3) placebo (normal saline). An in-plane ultrasound will be guide TAP blocks. Two subcostal injections will be applied by placing the probe midline and then moving lateral along the subcostal margin identifying area between the rectus abdominis sheath and the transversus abdominis muscle. The lateral two TAP block injections will be applied in the midaxillary line between the thoracic cage and iliac crest between external oblique and transversus abdominis muscles. Once the target area is positioned, the following injections will be given, based on randomization:

Liposomal bupivacaine. 40 ml of plain bupivacaine 0.25% will be mixed with 20 ml liposomal bupivacaine and 20 ml of saline. 20 ml of the mix will be injected at each location of the 4-quadrant TAP block.

Plain bupivacaine group. 50 ml of plain bupivacaine 0.5% will be combined with 30 ml of normal saline making a total of 80 ml. 20 ml will be injected at each location of the 4-quadrant TAP block.

Placebo group; patients will receive total of 80 ml of normal saline, injected 20 ml in each of the four-quadrant sites.

General anesthesia will be induced using propofol or etomidate, fentanyl, and rocuronium to facilitate intubation. Anesthesia will be maintained with sevoflurane or isoflurane, along with opioids and muscle relaxants as clinically indicated. However, intraoperative analgesic use will be limited to fentanyl, a short-acting opioid.

Postoperatively, patients will be given intravenous patient-controlled analgesia and nurses will be free to give additional opioid as clinically indicated. Hydromorphone will be the default drug, but fentanyl will be substituted if necessary. Clinicians blinded to trial drug will adjust analgesic management as necessary in an effort to keep verbal response pain scores (details below) <4 points on a 0-10 scale, with 10 being worst pain. When patients no longer need PCA, they will be switched to as-needed hydromorphone or fentanyl.

A single dose of dexamethasone (4-8 mg) will be permitted for PONV prophylaxis, and inhaled steroids will be permitted as necessary to treat reactive airway disease. The use of non-steroidal anti-inflammatory drugs and gabapentinoids will be allowed as part of the ERAS approach (enhanced recovery after surgery) according to hospital's clinical practice. Other opioid-sparing medications such as ketamine and lidocaine patches will not be permitted through the initial 72 postoperative hours.

Patients will be allowed to receive prophylactic anti-emetic (first choice ondansetron) intraoperatively based on the risk assessment for nausea and vomiting. Postoperative anti-emetics for symptomatic treatment will also be allowed; again ondansetron will be the first choice.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* 18-85 years old;
* ASA Physical Status 1-3;
* Scheduled for elective open or laparoscopic-assisted abdominal surgery;
* Anticipated hospitalization of at least three nights;
* Expected requirement for parenteral opioids for at least 72 hours for postoperative pain;
* Able to use IV PCA systems.

Exclusion Criteria:

* Hepatic disease, e.g. twice the normal levels of liver enzymes;
* Kidney disease, e.g. twice the normal level of serum creatinine;
* Bupivacaine sensitivity or known allergy;
* Women who are pregnant or breastfeeding;
* Anticoagulants considered to be a contraindication for TAP blocks;
* Surgeries with high port sites;
* Weight <50 kg.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Turan A, Ali Sakr Esa W, Brooker J, Rosen MJ, Ekrami E, Tok Cekmecelioglu B, Nair H, Al Jarkas A, Shah K, Mueller C, Valente M, El Hage Chehade N, Sessler DI; CLEVELAND Trial Group. Liposomal Bupivacaine, Plain Bupivacaine, and Saline for Transversus Abdominis Plane Blocks: The CLEVELAND Randomized Trial. Anesthesiology. 2026 Mar 1;144(3):546-558. doi: 10.1097/ALN.0000000000005869. Epub 2025 Dec 1. PMID 41329063

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine | Normal Saline
Started | 96 | 94 | 95
Completed | 89 | 84 | 88
Not Completed | 7 | 10 | 7

BASELINE CHARACTERISTICS:
Population: The analysis population is based on the modified intention to treat population comprising patients who completed the trial (261 patients total of 285).
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine | Normal Saline | Total
Number analyzed (Participants) | 89 | 84 | 88 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14) | 59 (13) | 59 (15) | 58 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 40 | 122
  Male | 46 | 45 | 48 | 139
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data on ethnicity was missing/not collected for some patients (n=1 in liposomal bupivacaine group, n=2 for plain bupivaacine group and n=4 for plain saline group)
  Participants
    Black: number analyzed (Participants) | 88 | 82 | 84 | 254
    Black | 9 | 8 | 9 | 26
    Hispanic: number analyzed (Participants) | 88 | 82 | 84 | 254
    Hispanic | 2 | 0 | 2 | 4
    Asian: number analyzed (Participants) | 88 | 82 | 84 | 254
    Asian | 1 | 0 | 1 | 2
    White: number analyzed (Participants) | 88 | 82 | 84 | 254
    White | 75 | 73 | 71 | 219
    Other: number analyzed (Participants) | 88 | 82 | 84 | 254
    Other | 1 | 1 | 1 | 3
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32 (6) | 31 (6) | 32 (6) | 32 (6)

OUTCOME MEASURES:

1. Primary Outcome: Total Opioids During Postoperative 24 Hours
Description: Opioid consumption, measured in morphine milligram equivalents, during the first 24 hours of surgery
Time Frame: Postoperative 24 hours
Population: Modified intention to treat population
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine | Normal Saline
Number analyzed (Participants) | 89 | 84 | 85
morphine milligram equivalents | 26 [18 to 48] | 33 [13 to 75] | 31 [17 to 53]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Normal Saline; Test type: Superiority; p = 0.355, Regression, Linear
Statistical Analysis 2: Comparison: Plain Bupivacaine vs Normal Saline; Test type: Superiority; p = 0.578, Regression, Linear

2. Primary Outcome: Total Opioid Consumption During Postoperative 24 to 48 Hours
Description: Total opioid consumption, in morphine milligram, equivalents, during postoperative 24 to 48 hours.
Time Frame: Postoperative 24 to 48 hours
Population: Modified intention to treat population
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine | Normal Saline
Number analyzed (Participants) | 89 | 84 | 88
morphine milligram equivalents | 10 [2 to 25] | 19 [5 to 42] | 15 [5 to 27]

3. Secondary Outcome: Time to Return of Sensation
Description: The investigator evaluate when patients feels both ice and pinprick in at least 6 of the 8 designated test locations, or 75% of the covered points if the TAP block did not initially cover all eight locations. The outcome is time (days) until sensation is recovered in 75% of the covered points.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine | Normal Saline
Number analyzed (Participants) | 79 | 73 | 83
days | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Normal Saline; Test type: Superiority; p = 0.248, Regression, Cox
Statistical Analysis 2: Comparison: Plain Bupivacaine vs Normal Saline; Test type: Superiority; p = 0.297, Regression, Cox

4. Secondary Outcome: Pain Scores During Postoperative 72 Hours
Description: Pain scores measured using the numeric rating scale (NRS) going from 0 to 10, with 0 representing least pain and 10 representing most pain.
Time Frame: Postoperative 72 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine | Normal Saline
Number analyzed (Participants) | 89 | 83 | 88
units on a scale | 4 [3 to 6] | 5 [3 to 6] | 4 [3 to 5]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Normal Saline; Test type: Superiority; p = 0.748, Mixed Models Analysis
Statistical Analysis 2: Comparison: Plain Bupivacaine vs Normal Saline; Test type: Superiority; p = 0.395, Mixed Models Analysis

5. Secondary Outcome: Total Opioid Consumption (Postoperative 48 to 72 Hours)
Description: Total opioid consumption, in morphine milligram equivalents, during postoperative 48 to 72 hours.
Time Frame: Postoperative 48 to 72 hours
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine | Normal Saline
Number analyzed (Participants) | 89 | 84 | 88
morphine milligram equivalents | 5 [0 to 15] | 9 [1 to 26] | 10 [0 to 18]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Normal Saline; Test type: Superiority; p = 0.152, Regression, Linear
Statistical Analysis 2: Comparison: Plain Bupivacaine vs Normal Saline; Test type: Superiority; p = 0.482, Regression, Linear

ADVERSE EVENTS:
Time Frame: Until discharge (approximately 5 days)
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/94 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/94 | 0/95
Other Adverse Events (participants affected / at risk) | 62/96 | 57/94 | 70/95
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Bupivacaine (N=96) | Plain Bupivacaine (N=94) | Normal Saline (N=95)
Opioid related side effects (General disorders) | 62 | 57 | 70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT04685876/Prot_SAP_000.pdf